CLINICAL TRIAL: NCT07352410
Title: Safety and Early Clinical Performance of High-Purity Type I Collagen Augmentation in Arthroscopic Meniscal Repair: A Prospective Feasibility Study
Brief Title: High-Purity Type I Collagen Augmentation in Meniscal Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIMS/IEC/006/2025
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Meniscus Tear; Knee Meniscus Injury; Meniscal Repair; Knee Arthroscopy (for Diagnostic or Therapy)
Keywords: Meniscal Tear; Meniscus Injuries; Knee Injuries; Arthroscopic Meniscal Repair; Meniscus Preservation; Biologic Augmentation; Collagen Scaffold; Type I Collagen; Cartilage Repair; Tissue Engineering
MeSH Terms: conditions — Knee Injuries; Osteogenesis Imperfecta, Type IV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-Purity Type I Collagen-Augmented Meniscal Repair (Experimental): Participants undergo standard arthroscopic meniscal repair augmented with High-Purity Type I Collagen applied at the repair site.
  Interventions: Device: High-Purity Type I Collagen

INTERVENTIONS:
Device: High-Purity Type I Collagen — Standard arthroscopic meniscal repair performed using established techniques (inside-out, outside-in, or all-inside). High-Purity Type I Collagen mesh is trimmed and applied over or within the repair site and secured using sutures or fibrin sealant, according to intra-operative requirements.

SUMMARY:
This prospective, single-arm feasibility study evaluates the safety, procedural feasibility, and early clinical outcomes of High-Purity Type I Collagen used as an adjunct in arthroscopic meniscal repair. The study aims to generate preliminary clinical, functional, and imaging data to inform the design of a future randomized controlled trial.

DETAILED DESCRIPTION:
Meniscal preservation is critical for long-term knee joint health, yet healing failure remains a concern, particularly in avascular zones. High-Purity Type I Collagen serves as a bioactive scaffold promoting cellular migration and early tissue integration. This study assesses early safety signals, feasibility metrics, patient-reported outcomes, and MRI-based healing characteristics following collagen-augmented meniscal repair.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years
* Symptomatic meniscal tear confirmed on MRI and indicated for arthroscopic repair
* Tear patterns amenable to repair
* Stable knee or concomitant ACL reconstruction permitted
* Ability to comply with rehabilitation and follow-up
* Written informed consent provided

Exclusion Criteria:

* Advanced knee osteoarthritis (Kellgren-Lawrence grade ≥3)
* Irreparable meniscal tears requiring meniscectomy
* Active joint infection or inflammatory arthritis
* Prior surgical repair of the index meniscus
* Known hypersensitivity to collagen products
* Systemic conditions impairing wound healing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety of High-Purity Type I Collagen Augmentation | From surgery to 2 months post-operatively
  Incidence of device-related adverse events, including infection, inflammatory reactions, synovitis, or need for re-operation.

SECONDARY OUTCOMES:
Pain Reduction Using Visual Analog Scale (VAS) | Baseline, 6 weeks, and 2 months
  Change in patient-reported knee pain measured using the Visual Analog Scale
Functional Outcome Using IKDC Subjective Knee Score | Baseline and 2 months
  Change in knee function assessed using the International Knee Documentation Committee (IKDC) subjective knee score.
Functional Outcome Using Lysholm Knee Score | Baseline and 2 months
  Assessment of knee stability and function using the Lysholm knee scoring system
Early Meniscal Healing on MRI | 2 months post-operatively
  MRI-based assessment of meniscal integrity, signal intensity at the repair site, and presence of fluid clefts or displacement
Objective Clinical Knee Examination Findings | Baseline, 6 weeks, and 2 months
  Assessment of knee effusion, range of motion, joint line tenderness, and meniscal provocation tests

CONTACTS AND LOCATIONS:
Overall Officials: Prema Dhanraj, MS, MCh, Study Chair — Rajarajeshwari Medical College and Hospital
Locations (1):
- Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
This feasibility study is exploratory in nature and not powered for hypothesis testing.

REFERENCES:
- [Background] Narayan N, Shivannaiah C, Gowda S. Evaluating the Efficacy of High-Purity Type I Collagen-Based Skin Substitute Versus Dehydrated Human Amnion/Chorion Membrane in the Treatment of Venous Leg Ulcers: A Randomized Controlled Clinical Trial. Cureus. 2025 Jul 30;17(7):e89031. doi: 10.7759/cureus.89031. eCollection 2025 Jul. PMID 40747200
- [Background] Narayan N, Gowda S, Shivannaiah C. A Randomized Controlled Clinical Trial Comparing the Use of High Purity Type-I Collagen-Based Skin Substitute vs. Dehydrated Human Amnion/Chorion Membrane in the Treatment of Diabetic Foot Ulcers. Cureus. 2024 Dec 5;16(12):e75182. doi: 10.7759/cureus.75182. eCollection 2024 Dec. PMID 39649230
- [Background] Bosisio FM, Estevez S. "Tire-bouchon" for vintage colloid. Int J Surg Pathol. 2013 Feb;21(1):47. doi: 10.1177/1066896912470163. No abstract available. PMID 23318609
- [Background] Paxton ES, Stock MV, Brophy RH. Meniscal repair versus partial meniscectomy: a systematic review comparing reoperation rates and clinical outcomes. Arthroscopy. 2011 Sep;27(9):1275-88. doi: 10.1016/j.arthro.2011.03.088. Epub 2011 Aug 6. PMID 21820843
- [Background] Lee HK, Yang Y, Su Z, Hyeon C, Lee TS, Lee HW, Kweon DH, Shin YK, Yoon TY. Dynamic Ca2+-dependent stimulation of vesicle fusion by membrane-anchored synaptotagmin 1. Science. 2010 May 7;328(5979):760-3. doi: 10.1126/science.1187722. PMID 20448186
- [Background] Duca RC, Hardy E, Salquebre G, Appenzeller BM. Hair decontamination procedure prior to multi-class pesticide analysis. Drug Test Anal. 2014 Jun;6 Suppl 1:55-66. doi: 10.1002/dta.1649. PMID 24817049
- [Background] Yamamoto H, Okumura S, Morita S, Obata K, Furuya K. Surgical correction of foot deformities after stroke. Clin Orthop Relat Res. 1992 Sep;(282):213-8. PMID 1516315
- [Background] Cleeland CS, Wang XS, Shi Q, Mendoza TR, Wright SL, Berry MD, Malveaux D, Shah PK, Gning I, Hofstetter WL, Putnam JB Jr, Vaporciyan AA. Automated symptom alerts reduce postoperative symptom severity after cancer surgery: a randomized controlled clinical trial. J Clin Oncol. 2011 Mar 10;29(8):994-1000. doi: 10.1200/JCO.2010.29.8315. Epub 2011 Jan 31. PMID 21282546